CLINICAL TRIAL: NCT06500325
Title: Results of Retrograde Titanium Elastic Nails for Fixation of Proximal Third Tibial Shaft Fractures in Children.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Youssery ahmed, Resident-Orthopedic surgery department-sohag hospital university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-20-06-12MS
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Proximal Third Tibial Shaft Fractures in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: retrograde titanium elastic nails for fixation of proximal third tibial shaft fractures in children — Two TENs were used in all cases using the double-C construct in most cases to gain three point of fixation. The starting point for nail insertion is 1.5-2.0 cm proximal to the physis of distal tibia. Both nails are then inserted through the entry holes and advanced to pass the level of the fracture site to achieve fixation. The two incisions for nail entry are closed in a layered fashion, and the wounds are well padded with gauze.

SUMMARY:
Pediatric tibial shaft fracture is the third most common pediatric long bone fracture after fracture of femur and forearm, representing 15% of all pediatric fractures. Closed reduction and casting is the standard of care for stable and minimally displaced fracture of the tibia in pediatric age group. Treatment of pediatric fractures dramatically changed in 1982. The goals are to stabilize the fracture, control limb length, alignment, rotation, instability, promote bone healing, and minimize the morbidity and complications for the child and his/her family. Titanium elastic nails (TENs) fixation was originally meant as an ideal treatment method for femoral shaft fractures, but was gradually applied to other long bones diaphysial fractures in children, as it represents a compromise between conservative and surgical therapeutic approaches with satisfactory results and minimal complications.

Over the past 20 years, pediatric orthopedic surgeons have tried a variety of methods to treat pediatric lower limb fractures to avoid prolonged immobilization and complications. Each method has had its own complications: cast immobilization alone or following traction had resulted in limb-length discrepancy, angulations, rotational deformity, psychological and economic complications. External fixation had resulted in pin-tract infection, loss of knee range of motion, delayed union, non-union, and refracture after fixator removal. TENs work by balancing the forces between the two opposing flexible implants. To achieve this balance, the nail diameter should be 40% of the narrowest canal diameter or more. The nails should assume a double-C construct. They should have similar smooth curve and same level entry points.

Ligier et al and Flynn et al have reported that TENs can give rotational stability if good care is taken intra-operatively during nail insertion and postoperatively, especially for comminuted, spiral, and long oblique fractures.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria included children are patients presented with traumatic proximal shaft tibia fracture closed or open up to Gustillo grade II and patients between 4 and 12.

Exclusion Criteria:

* Exclusion criteria excluded children presented with Gustillo grade III A, B & C open fractures and pathological fractures.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Goniometry of knee and ankle joints range of motion (ROM) | 1 year
  Goniometry involves using a goniometer, which is a specialized protractor-like device, to measure the angles of movement at joints such as the knee and ankle.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Patel NK, Horstman J, Kuester V, Sambandam S, Mounasamy V. Pediatric Tibial Shaft Fractures. Indian J Orthop. 2018 Sep-Oct;52(5):522-528. doi: 10.4103/ortho.IJOrtho_486_17. PMID 30237610
- [Background] Buechsenschuetz KE, Mehlman CT, Shaw KJ, Crawford AH, Immerman EB. Femoral shaft fractures in children: traction and casting versus elastic stable intramedullary nailing. J Trauma. 2002 Nov;53(5):914-21. doi: 10.1097/00005373-200211000-00017. PMID 12435943
- [Background] Ligier JN, Metaizeau JP, Prevot J, Lascombes P. Elastic stable intramedullary nailing of femoral shaft fractures in children. J Bone Joint Surg Br. 1988 Jan;70(1):74-7. doi: 10.1302/0301-620X.70B1.3339064.
- [Background] El-Adl G, Mostafa MF, Khalil MA, Enan A. Titanium elastic nail fixation for paediatric femoral and tibial fractures. Acta Orthop Belg. 2009 Aug;75(4):512-20. PMID 19774819